CLINICAL TRIAL: NCT01390987
Title: Survey Nazionale Sui Determinanti Del Ritardato Accesso Alle Cure e Della Mancata Aderenza al Trattamento Antitubercolare (National Survey on the Determinats of Delayed Access to Care and Non-adherence to Tuberculosis Treatment)
Brief Title: Access to Care and Adherence Tuberculosis (TB) Survey
Acronym: TBsurvey
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Giuseppe Lapadula, MD, PhD, Azienda Ospedaliera San Gerardo di Monza
Other Study IDs: TBsurvey-001
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prompt access to care and treatment adherence are the hearth of tuberculosis control.

This is a multicentre observational prospective study aimed at studying the factors associated with delayed access to care and low adherence to anti-tuberculosis treatment. Hetero- and self-administered questionnaires will be used at enrollment to assess clinical presentation and time and modalities of the diagnosis. Treatment adherence will be assessed during the follow-up with self administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 yrs of age
* recent new TB diagnosis
* Tuberculosis treatment prescribed
* Ability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All new tuberculosis (any site) diagnosed in the study time-frame, regardless of previous treatment history.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to TB diagnosis | Study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lapadula, MD, PhD, Principal Investigator — Clinic of Infectious Disease, AO San Gerardo, Monza, Italy
Locations (6):
- Italy (6):
  - AO Fallacara, Triggiano, BA
  - Clinic of Infectious Diseases, AO San Gerardo, Monza, MB
  - Clinica di Malattie Infettive, Spedali Civili, Brescia
  - Clinica di Malattie Infettive, Ospedale San Martino, Genova
  - Clinica di Malattie Infettive, Ospedale Luigi Sacco, Milan
  - Clinica di Malattie Infettive, Policlinico Gemelli, Roma

REFERENCES:
- [Derived] Peri AM, Bernasconi DP, Galizzi N, Matteelli A, Codecasa L, Giorgio V, Di Biagio A, Franzetti F, Cingolani A, Gori A, Lapadula G. Determinants of patient and health care services delays for tuberculosis diagnosis in Italy: a cross-sectional observational study. BMC Infect Dis. 2018 Dec 20;18(1):690. doi: 10.1186/s12879-018-3609-4. PMID 30572830